CLINICAL TRIAL: NCT02488603
Title: Utilization of Decision Aids for Tamoxifen Treatment in Breast Cancer Patients: A Randomized Controlled Trial.
Brief Title: Decision Aids for Tamoxifen Treatment in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Eun Sook Lee, MD, PhD, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: NCCKorea
Record Dates: First submitted 2015-06-25; First posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: Breast Neoplasms; Tamoxifen; Decision Aids
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques; Tamoxifen

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Decision aids (Experimental)
  Interventions: Behavioral: Decision aids (tamoxifen-related educational materials in brochure or mobile app); Drug: tamoxifen
- usual care (No Intervention)

INTERVENTIONS:
Behavioral: Decision aids (tamoxifen-related educational materials in brochure or mobile app) — Decision aids (tamoxifen-related educational materials in brochure or mobile app)
  Arms: Decision aids
Drug: tamoxifen
  Arms: Decision aids

SUMMARY:
This is an educational intervention study for breast cancer patients who undergo tamoxifen treatment. The purpose of the study is to assess the impact of decision aids (DA) on the patients' decision-making process, compliance on drug, and knowledge regarding tamoxifen treatment. Patients will randomly assign to DA group or conventional group. Both groups will have baseline questionnaire surveys before starting tamoxifen treatment, and 4 weeks later follow-up questionnaire surveys.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who are recommended to undergo tamoxifen treatment in National Cancer Center, Korea
* - Age at least 18 years and more

Exclusion Criteria:

* Age under 18 years
* Inability to read or speak Korean
* Disagree to provide a written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge of Tamoxifen Scale | baseline, 4weeks later

SECONDARY OUTCOMES:
Decisional Conflict Scale | baseline, 4weeks later
  Assess the decisional conflict regarding tamoxifen treatment
Satisfaction with Decision Questionnaire | baseline, 4weeks later
  Assess the satisfaction with decision to undergo tamoxifen treatment
EORTC QLQ-C30 Questionnaire | baseline, 4weeks later
  Assess the quality of life before and during tamoxfen treatment
EQ-5D Questionnaire | baseline, 4weeks later
  Assess the quality of life before and during tamoxfen treatment